CLINICAL TRIAL: NCT05950152
Title: A Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Analgesic Efficacy, Safety and Tolerability of Meloxicam Injection in Subjects After Abdominal Surgery
Brief Title: Efficacy, Safety and Tolerability Study of Meloxicam Injection in Subjects After Abdominal Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Collaborators: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLI-RD85-P2-2023
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Pain, Post-operative
MeSH Terms: conditions — Pain, Postoperative | interventions — Meloxicam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- meloxicam injection 30 mg (Experimental): meloxicam injection 30mg every 24 hours for up to 2 doses.
  Interventions: Drug: Meloxicam Injection 30mg
- meloxicam injection 60 mg (Experimental): meloxicam injection 60mg every 24 hours for up to 2 doses
  Interventions: Drug: Meloxicam Injection 60mg
- IV Placebo (Placebo Comparator): IV Placebo every 24 hours for up to 2 doses
  Interventions: Drug: Nacl 0.9%

INTERVENTIONS:
Drug: Meloxicam Injection 30mg — meloxicam injection 30mg every 24 hours for up to 2 dose
  Arms: meloxicam injection 30 mg
Drug: Meloxicam Injection 60mg — meloxicam injection 60mg every 24 hours for up to 2 dose
  Arms: meloxicam injection 60 mg
Drug: Nacl 0.9% — IV Placebo every 24 hours for up to 2 doses
  Arms: IV Placebo

SUMMARY:
The purpose of this study is to determine the analgesic efficacy and safety of Meloxicam Injection in subjects undergoing abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily provide written informed consent. Be scheduled to undergo elective abdominoplasty surgery without collateral procedures.

Be American Society of Anesthesiology (ASA) physical class 1 or 2. Male or female between 18 and 70 years of age, inclusive. Have a body mass index 18~30 kg/m2. Be able to understand the study procedures, comply with all study procedures, and agree to participate in the study program.

Exclusion Criteria:

Have a history of abdominoplasty surgery within the preceding 12 months. Have active or recent (within 6 months) gastrointestinal ulceration or bleeding.

Have a history of myocardial infarction or coronary artery bypass graft surgery within the preceding 12 months.

Have a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study.

Have a history of migraine or frequent headaches, seizures, or are currently taking anticonvulsants.

Have another painful physical condition that may confound the assessments of post operative pain.

Have a history of advanced malignant tumor. Have a history of alcohol abuse (regularly drinks > 4 units of alcohol per day; 8 oz. beer, 3 oz. wine, 1 oz. spirits) within the past 5 years or a history of prescription/illicit drug abuse.

Have positive results on the urine drug screen or alcohol breath test indicative of illicit drug or alcohol abuse.

Have evidence of a clinically significant 12 lead ECG abnormality. Have a clinically significant abnormal clinical laboratory test value. Have history of or positive test results for HIV, treponema pallidum,or hepatitis B or C.

Have a known allergy to meloxicam or any excipient of N1539, D5W, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs) or to any peri- or postoperative medications used in this study.

Have been receiving or have received chronic opioid therapy defined as greater than 15 morphine equivalents units per day for greater than 3 out of 7 days per week over a one-month period within 12 months of surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference Over the First 24 Hours (SPID24) | 24 Hours
  Pain intensity was recorded using a Numeric Pain Rating Scale (Range 0-10) where 0 equates to no pain (better), and 10 equates to the worst pain imaginable (worse). Pain intensity scores were to be recorded at the following time points: 0.25, 0.5, 0.75, 1, and 2 hours post Dose 1. Thereafter pain assessments were to be recorded every 2 hours until 48 hours post Dose 1. Pain intensity differences from baseline at each time point were calculated and a time weighted summed pain intensity difference (SPID) was then calculated. Time weighted SPID calculations were computed by multiplying a weight factor to each score prior to summation. The weight factor at each time point was the time elapsed since the previous observation. A smaller SPID value (i.e. more negative) was better.

SECONDARY OUTCOMES:
Summed Pain Intensity Difference (SPID) at Other Intervals | 48 Hours
  Pain intensity was recorded using a Numeric Pain Rating Scale (Range 0-10) where 0 equates to no pain (better), and 10 equates to the worst pain imaginable (worse). Pain intensity scores were to be recorded at the following time points: 0.25, 0.5, 0.75, 1, and 2 hours post Dose 1. Thereafter pain assessments were to be recorded every 2 hours until 48 hours post Dose 1. Pain intensity differences from baseline at each time point were calculated and a time weighted summed pain intensity difference (SPID) was then calculated. Time weighted SPID calculations were computed by multiplying a weight factor to each score prior to summation. The weight factor at each time point was the time elapsed since the previous observation. A smaller SPID value (i.e. more negative) was better.
Time to First Dose of Rescue Analgesia | 48 Hours
  Rescue analgesia (oral oxycodone 5 mg) was available to subjects with inadequately controlled pain upon request. Time to first rescue was calculated as the elapsed time from administration of Dose 1 to the administration of the first dose of rescue analgesia.
Number of Subjects Utilizing Rescue Analgesia | 48 Hours
  Rescue analgesia (oral oxycodone 5 mg) was available to subjects with inadequately controlled pain upon request.

CONTACTS AND LOCATIONS:
Locations (1):
- the Third XiangYa Medical Hospital of Central South University, Changsha, Hunan, China